CLINICAL TRIAL: NCT02577094
Title: Testing a Reduced Conditioning Regimen FB2A2 Preceded by a Fractionated Radio-immunotherapy (RIT) With 90Y-Epratuzumab Before Allogeneic Stem Cell Transplantation for Patients With Lymphocyte B CD22 Positive Acute Lymphoblastic Leukemia
Acronym: EPRALLO
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Gilead Sciences (Industry); Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC14_0429
Record Dates: First submitted 2015-10-02; First posted 2015-10-16 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Lymphocyte B CD22 Positive Acute Lymphoblastic Leukemia
Keywords: CD22 positive- lymphoblastic leukemia-RIT-Yttrium
MeSH Terms: interventions — Busulfan; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 90Y-DOTA-Epratuzumab IgG/Epratuzumab IgG — 2 injections of 90Y-DOTA- hLL2 IgG- hLL2 IgG at day -21 and day -14. (The 2 drugs are mixted in the same infusion)
  Other Names: 90Y-DOTA- hLL2 IgG and hLL2 IgG
Drug: Busulfan — Between the last injection of 90Y-DOTA- hLL2 IgG/hLL2 IgG (J-14) and the allogeneic stem cell transplantation
Biological: allogeneic stem cell transplantation. — At Day 0
Drug: Fludarabine — Between the last injection of 90Y-DOTA- hLL2 IgG/hLL2 IgG (J-14) and the allogeneic stem cell transplantation
Biological: Thymoglobulines — Between the last injection of 90Y-DOTA- hLL2 IgG/hLL2 IgG (J-14) and the allogeneic stem cell transplantation

SUMMARY:
Determination of the maximum tolerated dose (MTD) of fractionated RIT with epratuzumab radiolabeled with yttrium-90 (90Y-epratuzumab) preceding a reduced conditioning regimen FB2A2 before allogeneic stem cell transplantation.

DETAILED DESCRIPTION:
* Physical examination (screening and follow-up)
* Complete blood counts (screening and follow-up)
* Dosage of FLT3-ligand in plasma (screening and follow-up)
* Blood ionogramme, creatinine hepatic work-up (screening and follow-up)
* Left ventricular ejection fraction at pre-implant assessment
* Immunization test (screening and follow-up)
* Bone marrow aspiration or/and blood CD 22 immunophenotype for minimal residual disease evaluation (screening and follow-up)
* All exams which were initially abnormal and which are necessary for response evaluation and All exams which are needed in case of relapse suspicion.
* Pharmacokinetic of 90Y-hLL2

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Acute lymphoblastic Leukemia (ALL) CD22 + B-type in RC1 with high risk
* B-Cell Acute Lymphoblastic Leukemia (ALL) CD22+ beyond RC1.
* Expression of CD22 ≥ 30% in tumor population evaluated by flow cytometry or immunohistochemistry at diagnosis stage or relapse stage.
* HLA-identical donor intra family or not, without major HLA mismatch (9 / 10th accepted) without contra-indication for stem cell mobilization
* ECOG (Eastern Cooperative Oncology Group) ≤ 2
* Having or not received previously Epratuzumab
* Eligible for an allograft with reduced conditioning regimen
* With a signed informed consent
* Patient in age of children bearing with adequate contraception
* Patient affiliated to or beneficiary of the National Health Service

Exclusion Criteria:

* T-cell ALL
* Known hypersensibility to 90Y-DOTA-hLL2
* Immunization against hLL2 for patients having already received one or several injections of this antibody
* Patient eligible for myeloablative conditioning regimen
* Other prior malignancies must have had at least a 2-year disease-free interval with the exception of successfully treated carcinoma skin cancer or carcinoma in situ of the cervix.
* Patient with progressive psychiatric condition.
* HIV positive, hepatitis B-antigen positive, or hepatitis C positive patients who need a treatment
* Pregnant or breast-feeding women
* Women with childbearing potential without effective contraception
* Serious concomitant and uncontrolled infection
* Usual contraindications in the allogeneic transplant:
* Adult patient protected by the French law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Determination of the maximum tolerated dose (MTD) | 6 weeks
  Patient toxicity will be evaluated according to NTCAE V4 criteria.

SECONDARY OUTCOMES:
Overall survival | Month 12
Disease free survival at one year post-transplant | Month 12
Incidence of relapse at 1 year post-transplant | Month 12
Non relapse mortality at day 100 post-transplant | Day 100
Non relapse mortality at one year post-transplant | Month 12
Hematologic reconstitutions post-transplant | Month 3
  Biological follow-up
Immune reconstitutions post-transplant | Month 3
  Biological follow-up
Incidence of acute and chronic GVHD | Month 3 and 12
Chimerism post-transplant | Month 3
  Blood sample and/or bone marrow analysis by molecular biology
Residual disease post-transplant | Month 3 and Month 12
  by flow cytometry analysis
Toxicity of RIT | Week 6 and Month 12
  biological follow up and physical examination
Tolerance of RIT | Week 6 and Month 12
  biological follow up and physical examination
Immunization analysis : detection of antibody anti epratuzumab | Month 12
  By ELISA assay
90Y-DOTA-Epratuzumab blood pharmacokinetics | Month 2
  Detection of the radioactivity within the patient's blood samples
Dosage of FLT3-ligand in plasma and correlation with efficacy and toxicity of RIT | Month 12
  by biological assay